CLINICAL TRIAL: NCT01861951
Title: A Randomized Phase II Trial Comparing Pazopanib With Doxorubicin as First Line Treatment in Elderly Patients With Metastatic or Advanced Soft Tissue Sarcoma
Brief Title: A Trial Comparing Two Medications as First Treatment in Elderly Patients With Metastatic or Advanced Soft Tissue Sarcoma
Acronym: EPAZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Viktor Grünwald, Prof. , MD, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STS001; 2011-004168-30 (EudraCT Number)
Record Dates: First submitted 2013-04-11; First posted 2013-05-24 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2016-10

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; firstline treatment; eldery patients
MeSH Terms: conditions — Sarcoma | interventions — pazopanib; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pazopanib (Experimental): Pazopanib 800 mg, p.o., daily
  Duration of treatment:
  Until disease progression, treatment failure, or death due to any cause, whichever occurs first
  Interventions: Drug: Pazopanib
- Doxorubicin (Active Comparator): Doxorubicin 75 mg/m² BSA, d1, q3wk, i.v.
  Duration of treatment:
  Six cycles (approximately 18 weeks) or until disease progression, treatment failure, or death due to any cause, whichever occurs first
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Pazopanib
  Arms: Pazopanib
Drug: Doxorubicin
  Arms: Doxorubicin

SUMMARY:
Patients with a locally advanced or metastatic (i.e., there are already metastases of the diagnosed tumor in the body outside the primary lesion) soft tissue sarcoma will be recruited for this study. The minimum age to enter the study is 60 years.

Therapy with doxorubicin is the mainstay of palliative chemotherapy for these patients, which is associated with hematological toxicity and an increase of the infection rate. Pazopanib is known to rarely induce hematological toxicity or to trigger infection. We therefore assume that pazopanib exerts similar activity while decreasing neutropenia and neutropenic fever. Pazopanib is already approved in the U.S. and Europe for the treatment of advanced soft tissue sarcoma.

Doxorubicin and pazopanib will be randomly allocated to either receive doxorubicin or pazopanib in a phase II clinical trial. The aim of this study is to measure the treatment effect (reduction in tumor size or tumor stabilization) for both drugs, as well as the survival rate, and the duration of tumor control by the different therapies. A further objective is to measure the quality of life by standardized questionnaires throughout the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed written informed consent and willingness to comply with treatment and follow-up. Procedures conducted within 3 weeks as part of routine clinical management (e.g. blood count, imaging) and obtained prior to signing consent may be used for screening or baseline purposes if they are conducted as specified in the protocol
* 2. Male and female patients age ≥ 60 years at day of inclusion
* 3. Histologically confirmed diagnosis of metastatic or advanced soft tissue sarcoma of intermediate or high grade with disease progression within 6 months prior to study inclusion:

  * Fibrosarcoma
  * Pleomorphic high grade sarcoma ("malignant fibrous histiocytoma")
  * Leiomyosarcoma
  * Liposarcoma
  * Malignant glomus tumor
  * Rhabdomyosarcoma, alveolar or pleomorphic (excluding embryonal)
  * Vascular sarcoma (epithelioid hemangioendothelioma, angiosarcoma)
  * Synovial sarcoma
  * Not otherwise specified (NOS)
  * Malignant peripheral nerve sheath tumors
  * Other types of sarcoma (not listed as ineligible), if approved by the study coordinator.

Excluding:

Uncertain differentiation (epithelioid, alveolar soft part, clear cell, desmoplastic small round cell, malignant mesenchymoma, PEComa), chondrosarcoma, Ewing sarcomas/PNET, chordoma, malignant solitary fibrous tumors, embryonal rhabdomyosarcoma, osteosarcoma, gastrointestinal stromal tumors, dermatofibrosarcoma protuberans, inflammatory myofibroblastic sarcoma (low-grade), neuroblastoma, malignant mesothelioma, and mixed mesodermal tumors of the uterus (Study inclusion is based on local histopathological diagnosis).

* 4. ECOG performance status of 0-2
* 5. Evidence of progressive disease prior to start of treatment with measurable disease according to RECIST 1.1
* 6. Preferably archived tumor tissue of the most recent histology or, if not available, tumor block or 8 representative unstained sections on slides must be provided for all subjects for biomarker analysis within first month of treatment for central review
* 7. Adequate organ system function
* 8. Male patients with female partners of childbearing potential must meet one of the following criteria:

  * At least 6 weeks after surgical sterilization by vasectomy with documentation of azoospermia
  * Correct use of two reliable contraception methods for 14 days before exposure to IMP, through the dosing period, and for at least 21 days after the last dose of IMP. This includes every combination of a hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring) or an IUD/IUS with a barrier method (diaphragm, cervical cap, Lea contraceptive, femidom, or condom).
  * Complete sexual abstinence for 14 days before exposure to IMP, through the dosing period, and for at least 21 days after the last dose of IMP.
* 9. Female patients of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, as defined in Section "3.1 Inclusion criteria" during the study and for 14 days following the last dose of investigational product.

Exclusion Criteria:

* 1. Prior malignancy Excluding: Subjects who have had another malignancy and have been disease-free for 2 years, or subjects with a history of completely resected nonmelanomatous skin carcinoma, or successfully treated in situ carcinoma or incidental prostate cancer (TNM stage T1a or T1b) are eligible.
* 2. History or clinical evidence of CNS metastases Excluding: Subjects who have previously-treated CNS metastases (radiotherapy, surgery ± radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants 12 weeks prior to study inclusion. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases.
* 3. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including but not limited to:

  * Active peptide ulcer disease
  * Known intraluminal metastatic lesion(s) with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease) or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning of study treatment
* 4. Clinically significant gastrointestinal abnormalities that may affect absorption of IMP including but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowels
* 5. Presence of uncontrolled infection
* 6. QTc > 480 msecs using Bazett's formula
* 7. History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
* 8. Class III or IV congestive heart failure as defined by NYHA
* 9. Poorly controlled hypertension (SBP of ≤ 150 mmHg or DBP of ≤95 mmHg is acceptable provided that BP will be treated and monitored at least weekly. The goal is to attain controlled hypertension within 4 weeks of start of IMP which is defined as grade ≤1 hypertension CTCAE Version 4.0) Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed twice with an interval of at least

  1h before start of treatment and should be ≤140/90 mmHg for a subject to be eligible for the study. However, BP of ≤150/95 mmHg is acceptable provided the above measures are employed.
* 10. History of cerebrovascular accident including TIA, pulmonary embolism, or untreated DVT within the past 6 months Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
* 11. Major surgery or trauma within 28 days before first dose of IMP and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement are not considered to be major)
* 12. Evidence of active bleeding or bleeding diathesis
* 13. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* 14. Hemoptysis in excess of 2.5 mL once within 8 weeks of first dose of IMP
* 15. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* 16. Unable or unwilling to discontinue use of prohibited medications (see Section 5.5.5) for at least 14 days or 5 half-lives of a drug (whichever is longer) prior to the first dose of IMP and for the duration of the study
* 17. Treatment with any of the following anti-cancer therapies:

  * Radiation therapy, surgery, or tumor embolization within 14 days prior to the first dose of IMP OR
  * Chemotherapy, immunotherapy, biologic therapy, investigational therapy, or hormonal therapy within 14 days or 5 half-lives of a drug (whichever is longer) prior to the first dose of IMP 18. Any ongoing toxicity from prior anti-cancer therapy that is CTCAE > grade 1 and/or that is progressing in severity except alopecia
* 19. Prior systemic therapy for metastatic or advanced disease. Neoadjuvant or adjuvant chemotherapy is allowed, unless disease progression occurred within 6 months following end of treatment (see protocol chapter 5.4.2 for specifics)
* 20. Current participation in any other clinical trial and/or participation in another clinical trial within 30 days before the study begins
* 21. Known hypersensitivity to any component of IMPs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40 months | 10 to 40 months

SECONDARY OUTCOMES:
Change of rates of neutrophil granulocytopenia grade 4 (Day 1 - End of Trial (4 weeks after last IMP dose)), Change in rates of febrile neutropenia (Day 1 - End of Trial (4 weeks after last IMP dose)) | 10 months up to 40 months
Change from date randomization in progression-free rate at 12 weeks. Change from date randomization in progression-free rate at 26 weeks. | 10 months up to 40 months
Change from date of randomization in overall survival to date of death (from any cause) | 10 months up to 40 months
Change from date of randomization in objective response rate at 12 weeks. Change from date of randomization in objective response rate at 26 weeks. | 10 months up to 40 months
Collection of life quality questionnaires (QLQ-C30) at baseline, after 3, 6, 9, 12, 15, 19, and 26 weeks from date of randomization and end of therapy (EOT). Thereafter, assessment will be performed every 12 weeks until progression. | 10 months up to 40 months
Geriatric assessments from the date of baseline, after 12 and 26 weeks, and then every 12 weeks until progression | 10 months up to 40 months
Change in expression of certain biomarkers in blood to predict either response or resistance to pazopanib from baseline, week 2, day 1 of every cycle, week 19 and 26, end of therapy, and as part of the extension study every 6 weeks. | 10 months up to 40 months
Time from date of randomization until the date of first objective documentation of disease progression, treatment failure, or death due to any cause, whichever occurs first. | 10 months up to 40 months
Time to onset of response after 6, 12, 19 and 26 weeks from date of randomization | 10 months up to 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Gruenwald, MD, Prof., Principal Investigator — Hannover Medical School
Locations (11):
- University Hospitals Leuven, Leuven Cancer Institute, Dept. of General Medical Oncology, Leuven, Flemish Brabant, Belgium
- Germany (10):
  - Heidelberg University Hospital, Department of Internal Medicine, Hematology, Oncology and Rheumatology, Heidelberg, Baden-Wurttemberg
  - University Medical Centre Mannheim, Surgical oncology, Mannheim, Baden-Wurttemberg
  - Medical University Tuebingen, Center for Soft Tissue Sarcoma, GIST and Bone Tumors, Tübingen, Baden-Wurttemberg
  - LMU University hospital Munich Grosshadern, Medical Dept. III, Munich, Bavaria
  - Hannover Medical School, Department of Hematology, Hemostasis, Oncology and Stem Cell Transplantation, Hanover, Lower Saxony
  - University Hospital RWTH Aachen, Medical Dept. IV, Aachen, North Rhine-Westphalia
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - University Hospital Essen, West-German Tumor Center, Essen, North Rhine-Westphalia
  - University Hospital Carl Gustav Carus, Internal Medicine Dept. I, Dresden, Saxony
  - Charité Hospital, Medical Department, Division of Hematology, Oncology and Tumor Immunology, Berlin

REFERENCES:
- [Derived] Hamacher R, Liu X, Schuler MK, Hentschel L, Schoffski P, Kopp HG, Bauer S, Kasper B, Lindner L, Chemnitz JM, Crysandt M, Stein A, Steffen B, Richter S, Egerer G, Ivanyi P, Kunitz A, Grunwald V. A post hoc analysis of the EPAZ trial: The role of geriatric variables in elderly soft tissue sarcoma patients on toxicity and outcome. Eur J Cancer. 2023 Mar;181:145-154. doi: 10.1016/j.ejca.2022.12.012. Epub 2022 Dec 27. PMID 36657323
- [Derived] Grunwald V, Karch A, Schuler M, Schoffski P, Kopp HG, Bauer S, Kasper B, Lindner LH, Chemnitz JM, Crysandt M, Stein A, Steffen B, Richter S, Egerer G, Ivanyi P, Zimmermann S, Liu X, Kunitz A. Randomized Comparison of Pazopanib and Doxorubicin as First-Line Treatment in Patients With Metastatic Soft Tissue Sarcoma Age 60 Years or Older: Results of a German Intergroup Study. J Clin Oncol. 2020 Oct 20;38(30):3555-3564. doi: 10.1200/JCO.20.00714. Epub 2020 Aug 24. PMID 32840417
- [Derived] Crombie JL, Armand P. Diffuse Large B-Cell Lymphoma's New Genomics: The Bridge and the Chasm. J Clin Oncol. 2020 Oct 20;38(30):3565-3574. doi: 10.1200/JCO.20.01501. Epub 2020 Aug 19. No abstract available. PMID 32813609
- [Derived] Karch A, Koch A, Grunwald V. A phase II trial comparing pazopanib with doxorubicin as first-line treatment in elderly patients with metastatic or advanced soft tissue sarcoma (EPAZ): study protocol for a randomized controlled trial. Trials. 2016 Jul 7;17(1):312. doi: 10.1186/s13063-016-1434-x. PMID 27387325